CLINICAL TRIAL: NCT04541797
Title: Stress Cardiac Magnetic Resonance of Asymptomatic Type 2 Diabetics with Cardiovascular High Risk to Measure Empagliflozin Impact on Myocardial Blood Flow (CATCH-EM)
Acronym: CATCH-EM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: UW 19-010
Record Dates: First submitted 2020-07-08; First posted 2020-09-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes; Microvascular Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: double blinded randomised control trial study
Who Masked: Participant, Investigator
Masking Description: A stratified block randomisation process will be used. Two blocks will be created for randomisation which are 1) Positive stress CMR patients who did not have significant coronary artery disease; 2) Negative stress CMR patients. This will ensure equal spread of these two groups of patients into the control and intervention arm.
  Patients will be randomised into control and intervention arms. Control group: Patients will have placebo and optimised medical therapy and will continue to have protocol driven therapy and follow-up appointments (currently 1 appointment every 3 months).
  Intervention group: Patients will be prescribed empagliflozin 10mg once a day and optimised medical therapy for 6 months and standard follow-up like the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patients will have placebo and optimised medical therapy and will continue to have protocol driven therapy and follow-up appointments (currently 1 appointment every 3 months).
  Interventions: Drug: Placebo; Diagnostic Test: Stress Cardiac Magnetic Resonance
- Intervention (Experimental): Patients will be prescribed empagliflozin 10mg once a day and optimised medical therapy for 6 months and standard follow-up like the control group.
  Interventions: Drug: Empagliflozin 10 MG; Diagnostic Test: Stress Cardiac Magnetic Resonance

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Intervention group: Patients will be prescribed empagliflozin 10mg once a day and optimised medical therapy for 6 months and standard follow-up like the control group.
  Other Names: Empagliflozin
  Arms: Intervention
Drug: Placebo — Control group: Patients will have placebo and optimised medical therapy and will continue to have protocol driven therapy and follow-up appointments (currently 1 appointment every 3 months).
  Arms: Control
Diagnostic Test: Stress Cardiac Magnetic Resonance — Imaging: All patients will have stress CMR examinations at recruitment.
  Other Names: Stress CMR

SUMMARY:
The study design is a double blinded randomised control trial study that aims to conduct a randomised controlled trial of empagliflozin and determine if empagliflozin will improve myocardial blood flow in asymptomatic high risk type 2 diabetic patients. Also, to determine a cut-off using maximum upslope ratio and myocardial perfusion reserve index in which patients would demonstrate an improvement in myocardial blood flow.

DETAILED DESCRIPTION:
It is unknown whether empagliflozin will improve myocardial blood flow and resolve myocardial ischaemia caused by microvascular coronary artery disease in asymptomatic patients with type 2 diabetes.This study proposes to perform a randomised controlled trial to compare optimised medical therapy against empagliflozin in addition to optimised medical therapy to improve myocardial blood flow as measured by stress CMR. This trial would provide evidence if 10mg of empagliflozin given for 6 months could be an indicated treatment in asymptomatic high risk type 2 diabetic patients using stress CMR. The duration of 6 months is slightly longer than the mouse study (ie. 5 months) which showed an improvement in myocardial blood flow but not too long that the risk of increased patient withdrawal from the study will occur.

All patients will undergo coronary CT angiography in order to assess degree of coronary artery narrowing non-invasively before allocation to the control or intervention group. Patients will also undergo coronary CT angiography at the end of the study after 6 months of placebo or empagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Onset of type 2 diabetes at ≥30yrs old with no history of ketoacidosis
* 40-90yrs old
* Any 2 risk factors which include:

  i) Smoking (ie. current or ex-smokers) ii) Dyslipidaemia (defined as low density lipoprotein ≥2.6mmol/L, triglyceride >1.7mmol/L or decreased high density lipoprotein cholesterol <1.04mmol/L [man] or <1.29mmol/L [woman] or on lipid-lowering agent)(17, 18) iii) Hypertension (ie. systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg or patients treated for hypertension) iv) Obesity (using definition adapted for chinese ethnicity, body mass index >25kg/m2)(19) v) Family history of premature heart disease (defined as 1st degree relative [ie. parent or sibling] with development of atherosclerotic cardiovascular disease or cardiovascular related death <55 years of age in male and <65 years of age in female)
* HbA1c ≥ 6.5% and <10.0%

Exclusion Criteria:

* Angina pectoris or chest discomfort
* Prior coronary artery bypass grafts
* Coronary artery stenting within 6 months of study enrolment
* Previous myocardial infarct
* Any contraindication for stress CMR testing
* Renal impairment with eGFR <45ml/min/1.73m2
* Limited life expectancy <5 years, for example due to pulmonary disease, cancer or significant hepatic failure
* Contraindication to dual antiplatelet therapy
* Contraindication to empagliflozin or other SGLT2 inhibitors
* Unable to take empagliflozin
* Patients currently on empagliflozin or given empagliflozin in the last 6 months
* Planned need for concomitant cardiac surgery or coronary intervention
* Refusal or inability to sign an informed consent.
* Potential for non-compliance towards the requirements in the trial protocol (especially the medical treatment) or follow-up visits

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Difference in myocardial blood flow as measured by stress CMR (ie. maximum upslope ratio and myocardial perfusion reserve index) between patients receiving empagliflozin and patients not receiving empagliflozin. | 36 months
Cut-off value for maximum upslope ratio to predict ≥10% increase in myocardial blood flow as result of empagliflozin. | 36 months
Cut-off value for myocardial perfusion index to predict ≥10% increase in myocardial blood flow as result of empagliflozin. | 36 months
Changes in coronary artery plaque volumes between patients receiving empagliflozin and patients not receiving empagliflozin | 36 months

SECONDARY OUTCOMES:
Change in myocardial blood flow (MBF) in the intervention arm patients comparing patients with positive stress CMR to patients with negative stress CMR. | 36 months
Left ventricular ejection fraction. | 36 months
Left ventricular volumes. | 36 months
Left ventricular myocardial mass. | 36 months
Right ventricular ejection fraction. | 36 months
Right ventricular volumes. | 36 months
Right ventricular myocardial mass. | 36 months
Composite of empagliflozin therapy complication (eg. Urinary tract infection, acute renal failure). | 36 months
Progression in patient symptoms diagnoses. | 36 months
  The Seattle Angina Questionnaire (SAQ) will be administered at time of baseline CMR and at follow-up CMR in order to determine if there is an improvement in patient symptoms.
Improvement in exercise tolerance through performing a cardiopulmonary exercise test. | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong